CLINICAL TRIAL: NCT01196767
Title: Postoperative Analgesia After Cardiac Surgery: Effects of a Continuous Infusion of Ropivacaine Through Laterosternal Catheters
Brief Title: Ropivacaine Though Laterosternal Catheters After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHU-0080
Record Dates: First submitted 2010-07-26; First posted 2010-09-08 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Cardiac Surgery
Keywords: Sternotomy; Pain; Respiratory function; Opiates; Patient-controlled; Scheduled cardiac surgery under general anaesthesia without any locoregional anaesthesia protocol other than this presently studied
MeSH Terms: conditions — Pain; Respiratory Aspiration | interventions — Ropivacaine; Catheterization

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ropivacaine (Experimental)
  Interventions: Drug: Ropivacaine (in one arm); catheterization (in both).
- normal saline (Other)
  Interventions: Drug: Ropivacaine (in one arm); catheterization (in both).

INTERVENTIONS:
Drug: Ropivacaine (in one arm); catheterization (in both). — Parallel study with two groups:
  1. ropivacaine (2 mg.mL-1), at the rate of 4 mL.hr-1 through two subcutaneous catheters lateral to the sternum, both alimented by an elastomeric pump.
  2. same protocol, with normal saline instead of ropivacaine.

SUMMARY:
This is a prospective double-blinded and randomised study involving patients undergoing cardiac surgery with median sternotomy, the effects on postoperative analgesia of a 48-hr continuous infusion of ropivacaine 2 mg.mL-1, at the rate of 4 mL.hr-1 through two catheters inserted at the lateral edges of the sternum will be studied, versus a control group in which normal saline will be infused in the same conditions.

DETAILED DESCRIPTION:
Diverse methods for infusion of local anaesthetics after cardiac surgery have been proposed, but none of them provided high-level evidence of efficacy. The catheters studied here are designed for a surgical insertion before closure of the sternotomy, with the aim of infusing the drug the closest possible of the terminations of intercostal nerves.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled cardiac surgery.

Exclusion Criteria:

* - surgery in emergency
* thoracotomy
* cardiac graft
* redo
* pregnancy
* patient's refusal
* minor or adult under legal protection
* psychiatric ongoing disease
* addiction to opiates
* ongoing opiate treatment
* inability to use a PCA device
* respiratory insuffiency (Vital capacity or maximal expired volume per sec. < 50% of the expected value, or mean PAP > 50 mmHg)
* intra-aortic balloon
* severe renal insuffiency
* history of allergy or intolerance to: morphine, acetaminophen, bupivacaine.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pain score at mobilization (lying position for measurement of central venous pressure), expressed on a visual analogue scale. | every 4 hours during 48 hours

SECONDARY OUTCOMES:
Morphine consumption on PCA device | every 4 hours during 48 hours
Pain score at rest, expressed on a visual analogue scale. | every 4 hours during 48 hours
Vital capacity and inspiratory reserve volume, related to the preoperative values | daily during 48 hours
Postoperative blood level of troponin | every 8 hours during 48 hours
Arterial blood gases | every 4 hours during 48 hours
Time to first flatus | daily during 48 hours
Number of participants with adverse events | daily during 48 hours
  nausea and vomiting, pruritus
Postoperative blood level of ropivacaine at day + 1 and day + 2 | daily during 48 hours
Signs of intoxication to ropivacaine | eventual reports

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Eldjezi, MB, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Result] Eljezi V, Duale C, Azarnoush K, Skrzypczak Y, Sautou V, Pereira B, Tsokanis I, Schoeffler P. The analgesic effects of a bilateral sternal infusion of ropivacaine after cardiac surgery. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):166-74. doi: 10.1097/AAP.0b013e318240957f. PMID 22266899
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22266899